CLINICAL TRIAL: NCT03748342
Title: The Use of a Second-Generation Laryngeal Mask Airway Versus Endotracheal Tube in Obese Patients
Brief Title: Second Generation LMA Versus Endotracheal Tube in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Tiffany B Moon, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU-112017-050
Record Dates: First submitted 2018-10-22; First posted 2018-11-20 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Obese; Endotracheal Tube; Laryngeal Mask Airway
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Endotracheal Tube (No Intervention)
- Second-Generation LMA (Active Comparator)
  Interventions: Device: Second-Generation Laryngeal Mask Airway

INTERVENTIONS:
Device: Second-Generation Laryngeal Mask Airway — A second-generation LMA will be used for airway management (instead of ETT).
  Arms: Second-Generation LMA

SUMMARY:
This prospective, randomized, comparative study is intended to enroll a total of 148 patients with a BMI 30-49.9 kg/m2 undergoing surgery at Parkland Hospital. The efficacy and performance of a second-generation LMA will be compared to endotracheal intubation. A standardized anesthetic protocol that is usual and customary for the type of operation the patient is having will be provided to the anesthesia teams of enrolled subjects. The remainder of the anesthetic care of the subject will not deviate from the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Obese (BMI > or equal to 30 kg/m2
* Scheduled for a non-emergent surgery that requires general anesthesia (e.g., orthopedic, breast, urological, colorectal, ENT, vascular, general surgery)
* Willing and able to consent in English or Spanish
* No current history of advanced pulmonary or cardiac disease

Exclusion Criteria:

* Age less than 18 or older than 80
* BMI ≥50 or < 30 kg/m2
* Patient does not speak English or Spanish
* Expected surgical duration longer than 4 hours
* Planned postoperative ICU admission
* Patient refusal
* Monitored anesthesia care (MAC) or regional anesthesia planned
* Pregnant or nursing women
* "Stat" (emergent) cases
* Known or suspected difficult airway
* Full stomach/significant aspiration risk (gastroparesis, emergency surgery, untreated moderate to severe gastroesophageal reflux disease, hiatal hernia)
* No history of gastric surgery
* Surgery in position other than supine (e.g., Trendelenburg)
* Laparoscopic surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2025-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany S Moon, M.D., Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - Parkland Health & Hospital System, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Endotracheal Tube: Normal endotracheal tube
Period: Overall Study
Arm/Group | Standard Endotracheal Tube | Second-Generation LMA
Started | 48 | 49
Completed | 48 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Endotracheal Tube: 7.0/8.0 ETT
- Total: Total of all reporting groups
Arm/Group | Standard Endotracheal Tube | Second-Generation LMA | Total
Number analyzed (Participants) | 48 | 49 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.38 (13.63) | 47.06 (14.32) | 46.23 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 20 | 22 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 36 | 30 | 66
  Black | 5 | 14 | 19
  White | 7 | 5 | 12
BMI [Mean (Standard Deviation); unit: kg/m2] | 34.53 (4.91) | 35.8 (5.11) | 35.17 (5.03)
Smoking Status [Count of Participants; unit: Participants]
  Never | 34 | 34 | 68
  Used to but quit | 10 | 9 | 19
  Current Smoker | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Postoperative Hypoxia
Description: Patients in the 2 groups will be assessed for postoperative hypoxia (1 or more episodes) in the PACU using a visual analog scale.
Time Frame: Up to 80 minutes post-operatively
Measure: Number; unit: percentage of participants
Arm/Group | Standard Endotracheal Tube | Second-Generation LMA
Number analyzed (Participants) | 48 | 49
percentage of participants | 54.2 | 34.7

2. Secondary Outcome: Alterations in Blood Pressure
Description: Blood pressure monitor readings (events) will be recorded throughout the surgery and compared to baseline pre-operative values.
Time Frame: Intra-operatively
Measure: Number; unit: events
Arm/Group | Standard Endotracheal Tube | Second-Generation LMA
Number analyzed (Participants) | 48 | 49
events | 0 | 0

3. Secondary Outcome: Alterations in Heart Rate
Description: Heart rate monitor readings (events) will be recorded throughout the surgery and compared to baseline pre-operative values.
Time Frame: Intra-operatively
Measure: Number; unit: events
Arm/Group | Standard Endotracheal Tube | Second-Generation LMA
Number analyzed (Participants) | 48 | 49
events | 0 | 0

4. Secondary Outcome: Alterations in Oxygen Saturation (at Baseline)
Description: Oxygen saturation readings (events) will be recorded throughout the surgery and compared to baseline pre-operative values. Number of participants that did not require O2 is reported in the data table below.
Time Frame: Baseline
Measure: Number; unit: events
Groups:
- Standard Endotracheal Tube: Direct laryngoscopy performed and endotracheal tubeinserted.
Arm/Group | Standard Endotracheal Tube | Second-Generation LMA
Number analyzed (Participants) | 48 | 49
events | 0 | 0

5. Secondary Outcome: Alterations in Oxygen Saturation (at T15)
Description: Oxygen saturation readings (at T15- after 15 mins in PACU) will be recorded throughout the surgery and compared to baseline pre-operative values.
Time Frame: at 15 mins postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Endotracheal Tube | Second-Generation LMA
Number analyzed (Participants) | 48 | 49
Participants
  O2 required (SpO2<95%) | 10 | 10
  O2 not required | 38 | 39

6. Secondary Outcome: Alterations in Oxygen Saturation (at T45)
Description: Oxygen saturation readings (at T45- after 45 mins in PACU) will be recorded throughout the surgery and compared to baseline pre-operative values.
Time Frame: at 45 mins postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Endotracheal Tube | Second-Generation LMA
Number analyzed (Participants) | 48 | 49
Participants
  O2 required (SpO2<90%) | 3 | 0
  O2 required (SpO2<95%) | 3 | 3
  O2 not required | 42 | 46

7. Secondary Outcome: Alterations in Oxygen Saturation (at T80)
Description: Oxygen saturation readings (at T80- after 80 mins in PACU) will be recorded throughout the surgery and compared to baseline pre-operative values.
Time Frame: at 80 mins postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Endotracheal Tube | Second-Generation LMA
Number analyzed (Participants) | 47 | 49
Participants
  O2 required (SpO2<90%) | 3 | 0
  O2 required (SpO2<95%) | 2 | 1
  O2 not required | 42 | 48

8. Secondary Outcome: Alterations in Respiratory Rate
Description: Respiratory rate readings (events) will be recorded at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Standard Endotracheal Tube | Second-Generation LMA
Number analyzed (Participants) | 48 | 49
events | 16.33 (2.04) | 16.2 (2.16)

ADVERSE EVENTS:
Time Frame: until 1 hour after PACU arrival
Arm/Group | Standard Endotracheal Tube | Second-Generation LMA
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/49
Other Adverse Events (participants affected / at risk) | 0/48 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT03748342/Prot_SAP_000.pdf